CLINICAL TRIAL: NCT07347132
Title: Comparison of Pathological Outcome and Recurrence Rate Between En Bloc and Conventional Transurethral Resection of Bladder Tumor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lahore General Hospital (Other Government)
Responsible Party: Principal Investigator, Muhammad Irfan Jamil, Principal Investigator, Lahore General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LahoreGeneralH12
Record Dates: First submitted 2026-01-09; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Urinary Bladder Neoplasms; Non-muscle Invasive Bladder Cancer
Keywords: Transurethral Resection of Bladder Tumor; En Bloc Resection; Conventional Transurethral Resection; Tumor Recurrence
MeSH Terms: conditions — Urinary Bladder Neoplasms; Non-Muscle Invasive Bladder Neoplasms; Recurrence

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- En Bloc Transurethral Resection of Bladder Tumor (En Bloc TURBT) (Experimental): Participants were undergo complete removal of the bladder tumour as a single intact specimen (en bloc), including both exophytic and endophytic components, for tumours up to 1.5 cm in size.
  Interventions: Procedure: En Bloc Transurethral Resection of Bladder Tumor
- Conventional Transurethral Resection of Bladder Tumor (Conventional TURBT) (Active Comparator): Participants were undergo conventional piecemeal transurethral resection of the bladder tumour, in which the tumour is removed in multiple fragments.
  Interventions: Procedure: Conventional Transurethral Resection of Bladder Tumor

INTERVENTIONS:
Procedure: En Bloc Transurethral Resection of Bladder Tumor — Complete en bloc endoscopic resection of a non-muscle invasive bladder tumour (≤1.5 cm) as one piece, aiming to preserve specimen integrity and allow assessment of deep and lateral margins.
  Other Names: En bloc resection of bladder tumour (ERBT)
  Arms: En Bloc Transurethral Resection of Bladder Tumor (En Bloc TURBT)
Procedure: Conventional Transurethral Resection of Bladder Tumor — Piecemeal endoscopic resection of a non-muscle invasive bladder tumour by removing the lesion in multiple pieces, as per standard conventional technique.
  Other Names: Conventional transurethral resection of bladder tumour (cTURBT)
  Arms: Conventional Transurethral Resection of Bladder Tumor (Conventional TURBT)

SUMMARY:
Bladder cancer that has not invaded the bladder muscle often returns after treatment, creating repeated procedures and ongoing anxiety for patients. The standard initial treatment is transurethral resection of bladder tumour (TURBT), in which visible tumours are removed through a telescope passed into the bladder. Conventional TURBT usually removes the tumour in multiple pieces, which may reduce specimen quality for laboratory assessment and may increase the chance that small tumour fragments remain or spread during removal. En bloc TURBT is a newer technique that aims to remove the tumour in one intact piece, which may improve the quality of the tissue specimen for accurate staging and grading, allow better assessment of surgical margins, and potentially reduce recurrence.

This randomized controlled trial was conducted in the Department of Urology, Lahore General Hospital and PGMI, Lahore. A total of 116 adults (18 to 60 years) with non-muscle invasive bladder cancer were enrolled and randomly assigned to en bloc TURBT or conventional TURBT (58 patients per group). Resected specimens were evaluated by pathologists who was not be informed of the surgical technique. The study was compare key pathological outcomes, including the presence of detrusor muscle in the specimen, histological grade, tumour stage accuracy, specimen integrity, and the ability to assess lateral and deep resection margins. Participants were followed for 15 months, with surveillance at 3-month intervals.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female patients between 18 years and 60 years of age.
* Patients diagnosed with non-muscle invasive bladder cancer (NMIBC).
* Willingness to participate in the study, as indicated by signed informed consent.

Exclusion Criteria:

* Patients with muscle-invasive bladder cancer (MIBC) or metastatic disease.
* Previous history of bladder cancer treatment, including surgical resection or chemotherapy.
* Patients with contraindications to anesthesia or those unable to undergo TURBT due to medical reasons. iv. Individuals who have not provided informed consent or are unable to comply with follow-up requirements.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 116 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Tumor Recurrence Rate | Up to 15 months after surgery, assessed at 3, 6, 9, 12 and 15 months
  Proportion of participants with histologically confirmed recurrence of non-muscle invasive bladder cancer detected by cystoscopy and biopsy after complete initial resection.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Ijaz, Principal Investigator — Lahore General Hospital, Lahore
Locations (1):
- Lahore General Hospital, Lahore, Lahore, Punjab Province, Pakistan